## **Cover Page for ClinicalTrials.gov**

#### **Document:**

**Informed Consent Form** 

### **Official Study Title:**

Feasibility study of an adapted app-based anxiety intervention for autistic people.

#### **Document Date:**

January 05, 2023



# Feasibility study of an adapted app-based anxiety intervention for autistic people.

## Participant Consent Form

| Participant's Name:_ |
|----------------------|

| | Please initial |
|---|---|
| | if you agree |
| I confirm that I have read and understand the information sheet for this study, dated [insert relevant Version and date: Version XX, XX/XX/XXXX]. | , 3 |
| I have had the opportunity to consider the information and to ask questions. The research team have answered my questions satisfactorily. | |
| I understand that my participation is voluntary and that I am free to withdraw from the study at any time, without having to give any reason. This will not affect me, nor access to my usual health and social care services, in any way. I agree to the information I have already provided to be kept at the end of the study to make sure the research is reliable. | |
| I consent to the processing of my personal information and study data for the purposes explained to me in the information sheet. I understand that my information will be handled in accordance with European and local data protection laws. | |
| I understand and agree that my information may be subject to review by responsible individuals for monitoring and audit purposes. | |
| I agree for a notification letter to be sent to my GP so they are aware what the study involves for me. | |
| I understand that relevant sections of my medical notes may be looked at by the clinical research team, where it is relevant to this research. I give permission for the clinical research team to access to these records. | |
| I agree to install the Molehill Mountain app and to try to use the app daily for a 13-week period, to the extent that this is possible. I understand that I can use Molehill Mountain as much, or little, as I wish. | |
| I agree to participate in surveys about myself, my anxiety and personal goals, and my views of/ experiences using the Molehill Mountain app. This may be done via the secure Qualtrics online survey platforms, or in pen and paper format. | |
| Optional: I agree to take part in an interview about my views of/ experiences using the Molehill Mountain app. | |



| I agree for direct quotations from my optional interview to be used in publications, after any identifying information has been removed first. |
|---|
| I agree to the optional interview about my experiences of using the Molehill Mountain app being audio/ video recorded. |
| I agree to my Molehill Mountain app data being accessed by/ shared with the research team for the purposes of understanding how people are using the app, so that it can be improved in the future. |
| I understand there are legal obligations which might override confidentiality. Following local codes of ethics and conduct, researchers may breach confidentiality in exceptional circumstances where there is sufficient evidence that I may be a risk to my own, or others', safety. Researchers might also encourage me to seek support. |
| I consent to my study data being analysed and published. I understand that my confidentiality will be maintained and it will not be possible to identify me in any publication. |
| Optional: I consent to my completely anonymised data from this study being shared in the public domain for the purposes of open science and to support future research. |
| Optional: I consent to be contacted about future research projects. I will be able to decide then whether or not I want to participate in that study. |
| Optional: I would like to receive a copy of the results of the study once the research has ended. The research team might ask me for my feedback on the results, and I understand that this is completely optional. |



| Name of Volunteer: | | |
|--------------------------|---|-------|
| Signature of Volunteer: | | Date: |
| | • | |
| Name of Researcher: | | |
| Signature of Researcher: | | Date: |